CLINICAL TRIAL: NCT00697879
Title: A Phase I Study to Evaluate the Safety and Tolerability of the Histone Deacetylase Inhibitor, CHR-3996, in Patients With Advanced Solid Tumours
Brief Title: Safety Study of the Histone Deacetylase Inhibitor, CHR-3996, in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-3996-001; EudraCT Number: 2007-005043-19
Record Dates: First submitted 2008-06-10; First posted 2008-06-16 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Solid Tumor
Keywords: tumour; Solid tumour; histone deacetylase inhibitor; dose escalation; cancer
MeSH Terms: conditions — Neoplasms | interventions — 2-(6-(((6-fluoroquinolin-2-yl)methyl)amino)bicyclo(3.1.0)hex-3-yl)-N-hydroxypyrimidine-5-carboxamide; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Oral, once daily administration of CHR-3996 to determine safety and tolerability
  Interventions: Drug: CHR-3996

INTERVENTIONS:
Drug: CHR-3996 — Once daily oral ingestion of capsules (5, 10, 20 or 40 mg), dose depending on cohort, treatment cycle of 28 days
  Other Names: Histone deacetylase inhibitor; HDACi

SUMMARY:
CHR-3996 is one of a new class of anti-cancer agents - histone deacetylase inhibitors (HDACi) - that has exhibited pleiotropic activity both in vitro and in vivo against a range of human cancer cells. Regulation of the acetylation of both histone and non-histone proteins by histone deacetylase enzymes is one of the key mechanisms involved in epigenetic control of gene expression. HDACi have demonstrated activity in both in vitro cytotoxicity, and in vivo tumour xenograft studies

ELIGIBILITY:
INCLUSION CRITERIA:

1. Signed, informed consent
2. Histologically or cytologically confirmed malignant solid tumour refractory to standard therapy or for which no standard therapy exists
3. Recovered from all acute adverse effects of prior therapies (excluding alopecia and grade 1 neuropathy)
4. Adequate bone marrow, hepatic and renal function including the following

   1. Hb ≥ 9.0 g/dL, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥100 x 109/L
   2. Total bilirubin ≤ 1.5 x upper normal limit, excluding cases where elevated bilirubin can be attributed to Gilberts Syndrome
   3. AST (SGOT), ALT (SGPT) ≤ 2.5 x upper normal limit (or 5x UNL in the presence of liver metastases)
   4. Creatinine ≤ 1.5 x upper normal limit
5. Age ≥ 18 years
6. Performance status (PS) ≤ 2 (ECOG scale)
7. Estimated life expectancy greater than 3 months
8. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of trial. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception include IUD, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge)

EXCLUSION CRITERIA:

1. Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to trial entry (or a longer period depending on the defined characteristics of the agents used e.g. 6 weeks for mitomycin or nitrosourea, 3 months for antibodies). In patients with progressive disease, continuation of LHRH agonists for prostate cancer, bisphosphonates for bone disease and corticosteroids are permitted provided the dose does not change during the trial
2. Patients with a prior allogeneic haematopoietic stem cell transplant
3. Co-existing active infection or serious concurrent illness
4. Patients with significant cardiovascular disease as defined by:

   1. history of congestive heart failure requiring therapy
   2. history of angina pectoris requiring treatment or myocardial infarction within 6 months prior to trial entry
   3. presence of severe valvular heart disease
   4. presence of an atrial or ventricular arrhythmia requiring treatment
   5. LVEF below the normal range at the study centre
   6. Uncontrolled hypertension
   7. A history of QTc abnormalities or with a mean QTc interval >450 msec at screening
5. Any medical or other condition that in the investigator's opinion renders the patient unsuitable for this study due to unacceptable risk
6. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
7. Gastrointestinal disorders that may interfere with absorption of the study drug.
8. Patients with known brain tumours or metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
9. More than 6 prior chemotherapy regimens
10. Patients requiring growth factor support (erythropoietin, G(M)CSF, etc)
11. Patients requiring palliative radiotherapy within the last 4 weeks prior to study entry
12. Uncontrolled hypercalcaemia (>CTCAE v3 grade I)
13. Abnormal plasma potassium or magnesium levels (CTCAE v3 grade 3 or greater) despite therapy
14. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicities (DLT), maximum acceptable dose (MAD) and maximum tolerated dose (MTD) of CHR-3996 when administered orally to patients with advanced or treatment refractory solid tumours | After 28 days treatment

SECONDARY OUTCOMES:
To determine pharmacokinetic parameters of CHR-3996 | After 1 and 28 days treatment
To perform a preliminary assessment of the anti-tumour activity of CHR-3996 | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: F ALM Eskens, Dr, Principal Investigator — Erasmus MC University Medical Center; Udai Banerji, Dr, Principal Investigator — The Royal Marsden Hospital
Locations (3):
- Netherlands (2):
  - Erasmus MC University Medical Center - Location Centrum, Rotterdam
  - Erasmus University Medical Center - Location Daniel den Hoed, Rotterdam
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom